CLINICAL TRIAL: NCT00054041
Title: Phase II Evaluation Of SGN-00101 (HSP-E7) Fusion Protein In Women With Cervical Intraepithelial Neoplasia 3, CIN 3
Brief Title: Vaccine Therapy in Preventing Cervical Cancer in Patients With Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02513; GOG-0197; U10CA027469 (NIH); CDR0000269709 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia Grade 3; Human Papilloma Virus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

ARMS (2):
- Arm I (HspE7) (Experimental): Patients receive SGN-00101 subcutaneously once on weeks 1, 4, and 8 in the absence of disease progression. At week 15, all patients undergo large loop excision of the transformation zone under colposcopy.
  Interventions: Biological: HspE7; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Arm II (control) (Experimental): Patients receive standard care. At week 15, all patients undergo large loop excision of the transformation zone under colposcopy.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HspE7 — Given subcutaneously
  Other Names: HPV 16 E7/HSP65 Vaccine; HPV E7 Peptide Epitope Vaccine; SGN-00101
  Arms: Arm I (HspE7)
Procedure: therapeutic conventional surgery — Undergo large loop excision
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Vaccines made from antigens may make the body build an immune response to kill abnormal cervical cells and may be effective in preventing cervical cancer. Randomized phase II trial to study the effectiveness of vaccine therapy in preventing cervical cancer in patients who have cervical intraepithelial neoplasia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of SGN-00101, in terms of complete histologic regression, in patients with grade III cervical intraepithelial neoplasia.

II. Determine the toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine change in lesion size in these patients after treatment with this drug.

II. Compare histologic response before and after treatment with this drug in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive SGN-00101 subcutaneously once on weeks 1, 4, and 8 in the absence of disease progression.

Arm II: Patients receive standard care.

At week 15, all patients undergo large loop excision of the transformation zone under colposcopy.

Patients are followed at 19 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 28-84 patients (14-42 per treatment arm) will be accrued for this study within 12-48 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade III cervical intraepithelial neoplasia

  * Confirmed by biopsy or colposcopy
* Positive for human papilloma virus 16
* No endocervical glandular dysplasia
* No adenocarcinoma in situ
* Performance status - GOG 0-2
* No life-threatening or serious hematological disorder
* No life-threatening or serious hepatic disorder
* No life-threatening or serious renal disorder
* No life-threatening or serious cardiac disorder
* No life-threatening or serious respiratory disorder
* HIV negative
* Must be immunocompetent
* No history of autoimmune disease
* No life-threatening or serious immunological disorder
* No prior or concurrent severe allergic disease
* No concurrent human papilloma viral infection other than type 16
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No life-threatening or serious gastrointestinal disorder
* No life-threatening or serious endocrine disorder
* No invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No concurrent chronic or systemic steroids
* No prior organ transplantation
* No prior cancer therapy that would preclude study therapy

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-06; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Complete histologic regression of all CIN 3 lesions | Up to 3 years
  Fisher's exact test (and if feasible, Chi-Square test) will be conducted to see if the probability of responding in the investigational arm is significantly different from the controls actively accrued to this study. The conditional distribution used in Fisher's exact test will be used to calculate a 90% confidence interval for the odds ratio of observing a response in the investigational arm to the control arm.
Frequency and severity of adverse events assessed by Common Toxicity Criteria (CTC) version 2.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Trimble, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Roy AA, Pandey A, Dhas N, Hegde MM, Parekh HS, Andugulapati SB, Nandakumar K, Satish Rao BS, Mutalik S. The Confluence of Nanotechnology and Heat Shock Protein 70 in Pioneering Glioblastoma Multiforme Therapy: Forging Pathways Towards Precision Targeting and Transformation. Adv Pharmacol Pharm Sci. 2025 Apr 24;2025:1847197. doi: 10.1155/adpp/1847197. eCollection 2025. PMID 40313865